CLINICAL TRIAL: NCT06071624
Title: CD4CAR T Cell Therapy for CMML
Brief Title: Chimeric Antigen Receptor T Cell Therapy Redirected to CD4 (CD4CAR)as a Second Line Treatment for Chronic Myelomonocytic Leukemia, CMML.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huda Salman (Other)
Collaborators: iCell Gene Therapeutics (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor-Investigator, Huda Salman, Director, Hematologic Malignancies Service and Director, CAR T Cellular Therapy Program, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0840
Record Dates: First submitted 2023-09-15; First posted 2023-10-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia
Keywords: Chronic Myelomonocytic Leukemia; T Cell; Cell Therapy; CAR-T; chimeric antigen
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Redirected autologous T cells transduced with the anti-CD4 lentiviral vector (referred to as "CD4CAR" cells)
  Interventions: Biological: CD4CAR

INTERVENTIONS:
Biological: CD4CAR — CD4CAR cells transduced with a lentiviral vector to express the single-chain variable fragment (scFv) nucleotide sequence of the anti-CD4 molecule derived from humanized monoclonal ibalizumab and the intracellular domains of CD28 and 4-1BB co-activators fused to the CD3ζ T-cell activation signaling domain administered by IV infusions as a single dose

SUMMARY:
This study is designed as a single arm open label traditional Phase I, 3+3, study of CD4-directed chimeric antigen receptor engineered T-cells (CD4CAR) in patients with relapsed or refractory CMML. Specifically, the study will evaluate the safety and feasibility of CD4CAR T-cells.

DETAILED DESCRIPTION:
The study will be performed as a dose-escalation protocol. Due to the relatively low incidence and prevalence of cluster of differentiation 4-positive (CD4+) hematological malignancies and the associated aggressive nature of these diseases and the sequel of treatment failure, the investigators expect to recruit 20 subjects at Indiana University with an expected dropout rate of 25% primarily due to rapid progression or death and screen and or manufacturing failure. Taking this into account, the investigators expect to treat 15 patients. The study will utilize autologous CD4CAR T-cells that are engineered to express a chimeric antigen receptor (CAR) targeting CD4 that is linked to the cluster of differentiation 28 (CD28), 4-1BB, cluster of differentiation 3-zeta (CD3ζ) signaling chains (third generation CAR).

At entry, disease status will be staged. Qualifying subjects will be leukapheresed to obtain large numbers of peripheral blood mononuclear cells (PBMC) for the manufacturing. Next, participants will receive conditioning chemotherapy. If tumor burden is sufficiently reduced (screening step), participants will receive CD4CAR cells by infusion on Day 0 of treatment.

If the disease progresses during the manufacturing period participants may be excluded from the study. Minimal chemotherapy to keep the disease under control in the meanwhile is allowed if deemed necessary by investigators.

A single dose of CD4CAR transduced T cells will consist of the cell number for the dose level to be infused.

Post-infusion monitoring of CD4CAR T-cells: Subjects will have blood drawn for cytokine levels, CD4CAR Transgene Copy Number (PCR) and flow cytometry in order to evaluate the presence of CD4CAR cells on days 0, 1, 3, 5, 7, 14, and 28 following infusion (or as clinically needed). Cytokines levels will be evaluated per schedule above in addition to and as needed every 8 +/- 2 hours as feasible if/when CRS occurs and until resolution. Active monitoring of fungal and viral infections during treatment while utilizing standard prophylaxis recommended for HIV-positive patients with T-cell aplasia and those undergoing allogeneic stem cell transplant. Investigators plan to collect data about clinicoradiologic measurements of residual tumor burden starting on day 7 and weekly afterward until Day 28 and then monthly for 6 months. This will be followed by quarterly clinical evaluations for the next two (2) years with a medical history, physical examination, and comprehensive blood testing. After these short- and intermediate-term evaluations are performed, these patients will enter a rollover study to assess for disease-free survival (DFS), relapse, and the development of other health problems or malignancies where follow-up will be up to twice a year by phone and a questionnaire for an additional thirteen (13) years. The treating physician will decide to proceed with allogeneic or autologous transplant when needed.

Dose of CD4CAR description: the main objective of this study is to establish a recommended dose and/or schedule of CD4CAR. The guiding principle for dose escalation in phase I is to avoid unnecessary exposure of patients to sub-therapeutic doses (i.e., to treat as many patients as possible within the therapeutic dose range) while preserving safety and maintaining rapid accrual. Investigators will use the rule-based traditional Phase I "3+3" design for the evaluation of safety. Based on lab experience in mice the starting dose (dose level 1) for the first cohort of three patients in phase I portion of the study will be 8x10^5 cells. The dose escalation or de-escalation will follow a modified Fibonacci sequence as below.

If more than one patient out of the first cohort of three patients in dose level 1 experience dose limiting toxicity (DLT), the trial will be placed on hold. If zero or one out of three patients in the first cohort of dose level 1 experience DLT, three more patients will be enrolled at dose level 1; the dose escalation continues until at least two patients among a cohort of six patients experience DLT (i.e., ≥33% of patients with a DLT at this dose level)

If one of the first three patients in dose level 1 experiences a DLT, three more patients will be treated at dose level 1.

If none of the three patients or only one of the 6 patients in the dose level 1 experiences a DLT, the dose escalation continues to the dose level 2 If one of the first three patients in dose level 2 experience a DLT, three more patients will be treated at dose level 2 If none of the three patients or only one of the 6 patients in the dose level2 experiences a DLT, the dose escalation continues to the dose level 3 If one of the first three patients in dose level 3 experiences a DLT, three more patients will be treated at dose level 3 If none of the three patients or only one of the 6 patients in the dose level 3 experiences a DLT, dose level 3 will be declared the maximum tolerated dose (MTD) and will be used as the recommended phase II dose (RP2D) for the phase II portion of the study.

In summary, the dose escalation continues until at least two patients among a cohort of six patients experience DLT (i.e., ≥33% of patients with a DLT at that dose level). The recommended dose for phase II trials is defined as one dose level below this toxic dose level. Since some grade 3 and possibly 4 toxicities are highly likely to be reversible, grade 3 infectious, hematological and vascular toxicities will not be considered DLTs mandating dose reduction. Also allergic or infusion-related reactions ≤ grade 3 will not be counted as DLTs. There will be no intra-patient dose escalation or reduction.

To allow for full spectrum toxicity duration evaluation and reporting, no patients within the same or a different cohort will be initiated on lymphodepleting chemotherapy sooner than 28 days from the initiation date of the preceding patient.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Diagnosis of CMML that is CD4+ and is recurrent or refractory to first line standard of care treatment.
4. Creatinine clearance of ≥ 60 ml/min (or otherwise non clinically significant, per study investigator)
5. ALT/AST < 3 x ULN
6. Bilirubin < 2 x ULN
7. Pulmonary Function Test (PFT) with a DLCO of ≥ 50%. This will not have to be repeated if within 45 days of initial assessment.
8. Adequate echocardiogram with EF of ≥50% This will not have to be repeated if within 45 days of initial assessment.
9. Adequate venous access for apheresis and no other contraindications for leukapheresis

Exclusion Criteria:

1. CD4 negative CMML
2. Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential (see definition below) must have a negative serum or urine pregnancy test prior to initiation of conditioning chemotherapy, per research sites' clinical policy
3. Uncontrolled active infection necessitating systemic therapy
4. Active hepatitis B or hepatitis C infection. Active hepatitis C is defined as the hepatitis C antibody is positive while quantitative HCV RNA results exceed the lower detection limit

   Note the following subjects will be eligible:
   * Subjects with a history of hepatitis B but have received antiviral therapy and have non-detectable viral DNA for 6 months prior to enrollment are eligible
   * Subjects seropositive for HBS antibodies due to hepatitis B virus vaccine with no signs or active infection (Negative HBs Ag, HBc and HBe Ags) are eligible
   * Subjects who had hepatitis C but have received antiviral therapy and show no detectable hepatitis C virus (HCV) viral RNA for 6 months are eligible
   * If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative
5. Concurrent use of systemic glucocorticoids in greater than replacement doses or steroid dependency defined in rheumatological and pulmonary diseases as uninterrupted corticosteroid intake for more than a year at a dosage of 0.3 mg/kg/day or greater, and where the underlying disease worsens on temporary stoppage of steroid therapy, with symptoms of steroids withdrawal (eg, lethargy, headache, weakness, pseudo rheumatism, emotional disturbances, etc) precipitated by the temporary stoppage unless tapering can occur safely without compromising the underlying disease, the withdrawal tolerance and can happen in a timeframe appropriate to enroll in this trial without safety concerns

   Subjects who receive daily corticosteroids in replacement doses can be included in the study. The replacement doses are defined as following:
   1. Hydrocortisone 25mg/day or less
   2. Prednisone 10mg/day or less
   3. Dexamethasone 4mg or less - Note: Recent or current use of inhaled glucocorticoids is not exclusionary, as this route pertains extremely minimal systemic penetration
6. Any previous treatment with any gene therapy products
7. Any uncontrolled active medical disorder that would preclude participation as outlined in the opinion of the treating investigator and/or Principal Investigator
8. HIV infection
9. Subjects who have received or will receive live vaccines within 30 days before the first experimental cell treatment. Inactivated seasonal flu vaccination is allowed
10. Subjects with active autoimmune diseases who need systematic treatments (such as disease modifying agents, corticosteroids and immunosuppressive drugs) during the last year Note: Replacement therapy (thyroxine, insulin or physiological corticosteroid replacement therapy (up to10 mg of oral daily prednisone or equivalent in hydrocortisone and dexamethasone) to treat adrenal dysfunction or pituitary dysfunction) is not considered as systematic therapy. Subjects who need inhalation corticosteroid therapy can be included in this trial. Subjects with vitiligo or in long-term remission of pediatric asthma or allergic diseases can be included in this trial
11. Subjects with a history of mental disorders or drug abuse that may influence treatment compliance
12. Active malignancy not related to CMML that has required therapy in the last 3 years or is not in complete remission. Exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy. Other similar malignant conditions may be discussed with and permitted by the Principal Investigator
13. Participation in a cell/gene therapy clinical study with an investigational product within the past 6 months; and/or no other clinical trial with an investigational product within the last 4 weeks, provided subject was in fact given that experimental treatment, just being enrolled and treated is not a disqualifier.

Eligibility for cd4CAR Infusion

1. Afebrile and not receiving antipyretics, and no evidence of active infection. If fever is attributed to underlying disease, it will not disqualify.
2. Specific organ function criteria for cardiac, renal, and liver function must be similar to initial inclusion values. Tests such as echocardiogram and PFTs need not be repeated if within 45 days of initial assessment
3. If previous history of corticosteroid chemotherapy, subject must be off all but adrenal replacement doses 3 days before the CD4CAR infusion
4. Planned infusion dose was successfully manufactured and met release criteria

5.5 Contraception and Reproductive Potential Guidelines

Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test prior to conditioning chemotherapy.

Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double barrier methods of contraception from time of consent through at least 90 days after CD4CAR infusion.

Acceptable birth control includes a combination of two of the following methods:

* Condoms (male or female) with or without a spermicidal agent.
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormonal-based contraception

Subjects who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy, salpingotomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception. Acceptable documentation of sterilization, azoospermia, and menopause is specified next:

Written or oral documentation communicated by clinician or clinician's staff of one of the following:

* Physician report/letter
* Operative report or other source documentation in the subject record (a laboratory report of azoospermia is required to document successful vasectomy)
* Discharge summary
* Laboratory report of azoospermia
* Follicle stimulating hormone measurement elevated into the menopausal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
Dose finding: Maximum tolerated dose (MTD) is defined as one dose level lower than the dose limiting toxicity (DLT) of the CD4CAR in CMML | Day 0 through Day 28 post-infusion
  In this traditional phase 1 dose escalation, cohorts of three subjects will be treated on a dose level that will be incremented to next dose level if no dose limiting toxicities (DLT) were reported or expanded if a DLT is documented
The efficacy of treatment with CD4CAR and description of CMML response to CD4CAR | Day 28 through 6 months post-infusion
  serial marrow sampling will be analysed for response as measured by reduction on the CMML clonal cells at different time points. Other measures include reduction on transfusion dependency and molecular remissions if at diagnoosis molecular markers were identified.

SECONDARY OUTCOMES:
in vivo persistence of a single dose of the CD4CAR in patients with CMML | Day 0 through Day 28
  Flowcytometry and transgene copy number by PCR will be used to evaluate the CAR T cell persistence post infusion
efficiacy of the CD4CAR to target T regulatory cells and myeloid derived suppressor cells | Day 0 through Day 28 post-infusion
  T regs estimation in marrows will be done at diagnosis and on Day 28 post-infusion. This will be done by flowcytometry to assess the reduction on these cells phenotyped by double positivity for CD4 and FOXP3. At the same time points Myeloid Derived Suppressor Cells (MDSCs), will also be quantified. MDSCs will be identified by a master mix of commercially available antibodies against MDSC subsets including CD16, CD15, CD14, CD45, CD84.etc, Cytek® cFluor® MDSC Ki panel.

CONTACTS AND LOCATIONS:
Overall Officials: Huda Salman, MD, PhD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida 33136, Miami, Florida
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Albert Einstein Health Network, The Bronx, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas